CLINICAL TRIAL: NCT06873360
Title: Design of a Medical Device for Oxaliplatin-Induced Peripheral Neuropathy Considering the Patient's Voice in Gastrointestinal Cancer
Brief Title: Medical Device for Oxaliplatin-Induced Neuropathy in Gastrointestinal Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Sandra Soriano-Sánchez, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: 2024/5114
Record Dates: First submitted 2025-02-15; First posted 2025-03-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy
Keywords: Peripheral Neuropathy Induced by Oxaliplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group of patients with gastrointestinal cancer treated with oxaliplatin.
  Interventions: Other: Clinical interviews with patients and Usability interviews and glove testing.

INTERVENTIONS:
Other: Clinical interviews with patients and Usability interviews and glove testing. — Clinical interviews with patients: These will be conducted by nursing staff with an approximate total of 50 patients during their treatment at the Hospital. Each interview will last 15 minutes. Under no circumstances will the patient be required to answer any question.
  Usability interviews and glove testing: 10 patients selected from the previous interviews will test different gloves with various textures and levels of stiffness. Additionally, other questions will be asked focusing on refining the design. This evaluation will help determine the most suitable materials for the device's manufacturing, achieving a balance between comfort, discretion and functionality.

SUMMARY:
This is an observational study related to a medical device designed for the prevention of oxaliplatin-induced peripheral neuropathy (OIPN) in patients with gastrointestinal cancer. The primary objective is to collect data through interviews with patients experiencing OIPN symptoms to co-design the medical device prototype, incorporating the patient's perspective. Additionally, the study aims to identify clinical and usability patterns that will help optimize the design of a future clinical investigation assessing the safety and efficacy of the final device.

DETAILED DESCRIPTION:
Main Hypothesis:

The clinical data collected from patient interviews, along with their active participation in the co-design of the localized cooling medical device, likely in the form of gloves, will enable the design of both the functional prototype and the future clinical research on safety and efficacy. This approach will increase the likelihood of patient acceptance of the medical device treatment and help identify different patient profiles that could benefit the most from it.

Secondary Hypotheses:

1. Patients will be able to easily adhere to the use of the device during chemotherapy.
2. The final glove design, in terms of materials and structure, will be suitable for commercial manufacturing and will have a viable demand among patients and healthcare providers.
3. There is no difference in treatment adherence between men and women or among people of different ages.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient patient with gastrointestinal cancer treated with oxaliplatin.
* Having completed at least three cycles of chemotherapy.
* Presenting acute or chronic symptoms of chemotherapy-induced peripheral neuropathy.
* The study will include individuals over 18 years old. Gender identify will be collected confidentially and inclusively, offering options for non-binary individuals and those who prefer not to identify with binary categories.

Exclusion Criteria:

* Patient with osteoarthritis or arthritis in the hands.
* Diagnosis of any autoimmune disease affecting connective tissue, such as: rheumatoid arthritis, Raynaud's syndrome, lupus, scleroderma, dermatomyositis, vasculitis, or cryoglobulinemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal cancer treated with oxaliplatin chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Co-design a medical device with patients to develop a solution that can prevent the onset of oxaliplatin-induced peripheral neuropathy (OIPN) | From baseline to 6 months
  Interviews will be conducted with patients to gather information on the clinical presentation of oxaliplatin-induced peripheral neuropathy and its impact on patients' quality of life.

SECONDARY OUTCOMES:
Gain an in-depth understanding of the progression of OIPN symptoms. | From baseline to 6 months
  It consists of understanding the evolution of symptoms of oxaliplatin-induced peripheral neuropathy through quality of life questionnaires. These quality of life questionnaires will include questions related to intensity, location, triggers, and recurrence of these symptoms.
Ensure the usability of the device by assessing the patient's ability to adhere to treatment with a medical device. | From baseline to 6 months
  The patients will try different gloves with various textures and levels of stiffness. Additionally, other questions different from those in the main study will be asked, focusing more on refining the design. This evaluation will help determine the most suitable materials for the device's manufacturing, achieving a balance between comfort, discretion, and functionality.
Determine the design characteristics of the gloves. | From baseline to 6 months
  The patients will receive three different designs of non-functional commercial gloves (which do not generate cold or heat through electronics). In some cases, these gloves may have been modified to exhibit certain properties (such as texture, breathability, or thickness). Additionally, different sizes will be available for each model to ensure a proper fit for the patient's hand.

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain